CLINICAL TRIAL: NCT02872220
Title: A Randomized Study to Assess the Potential for Photoallergy of SPF 50 Y65 110, SPF 50 Y51 002 and SPF 15 V27 104 in Human Subjects
Brief Title: To Test for Photo Allergy Reaction of Sunscreens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 18291
Record Dates: First submitted 2016-06-14; First posted 2016-08-19 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Photoallergy
MeSH Terms: conditions — Dermatitis, Photoallergic | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SPF 50 Y65 110, SPF 50 Y51 002, and SPF 15 V27 104 (Experimental): All test products compared to that of a negative control [0.9% NaCl] were tested simultaneously on each subject.
  Interventions: Drug: SPF 50 Y65 110 (BAY987519); Drug: SPF 50 Y51 002 (BAY987519); Drug: SPF 15 V27 104 (BAY987519); Drug: Sodium chloride [NaCl]

INTERVENTIONS:
Drug: SPF 50 Y65 110 (BAY987519) — Application of 200 µL in an occlusive patch of Webril (0.150 ± 0.010 mg) compared to that of a negative control (0.9% sodium chloride, NaCl) and followed by irradiation with UV A and UVB.
Drug: SPF 50 Y51 002 (BAY987519) — Application of 200 µL in an occlusive patch of Webril compared to that of a negative control (0.9% sodium chloride, NaCl) and followed by irradiation with UV A and UVB.
Drug: SPF 15 V27 104 (BAY987519) — Application of 200 µL in an occlusive patch of Webril compared to that of a negative control (0.9% sodium chloride, NaCl) and followed by irradiation with UV A and UVB.
Drug: Sodium chloride [NaCl] — Negative control (200 µL, 0.9% sodium chloride [NaCl]) after a single 24 h application of test materials followed by irradiation with ultraviolet A (UVA) and ultraviolet B (UVB).

SUMMARY:
The primary objective of this tudy was to evaluate the potential of photoallergy of of sun care products Sun Protection Factor (SPF) 50 Y65 110, SPF 50 Y51 002, and SPF 15 V27 104 application compared to that of a negative control (0.9% sodium chloride, NaCl) and followed by irradiation with UV A and UVB.

The secondary objective aims for evaluation of the safety of SPF 50 Y65 110, SPF 50 Y51 002, and SPF 15 V27 104 combined with ultraviolet (UV) A/B irradiation by monitoring adverse events (AEs) throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, aged 18 to 65 with good general health
* Fitzpatrick skin type I IV
* Females (of childbearing potential) on acceptable measure of contraception
* Willing to follow study rules, which include: no sun exposure (for example, no swimming, sunbathing, or tanning beds), avoidance of activities that would cause excessive sweating, no use of lotions, creams, or oils on the back area
* Willing to not change the current brand of personal care products such as soaps, body washes, laundry detergent, body sprays, body spritzes, etc. while participating in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-03-23 (Actual); Primary Completion 2015-05-08 (Actual); Study Completion 2015-05-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of inflammatory responses | up to 3 weeks
  Inflammatory responses (Based on scores): 0 = No visible reaction + = Slight, confluent, or patchy erythema 1 = Mild erythema (pink) 2 = Moderate erythema (definite redness) 3 = Strong erythema (very intense redness)
Evaluation of superficial effects | up to 3 weeks
  Superficial effects: g = Glazing y = Peeling c = Scab, dried film of serous exudate of vesicular or bulla reaction d = Hyperpigmentation (reddish brown discoloration of test site) h = Hypopigmentation (loss of visible pigmentation at test site) f = Fissuring grooves in the superficial layers of the skin

SECONDARY OUTCOMES:
Adverse event collection as a measure of safety and tolerability | up to 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Pinellas Park, Florida, United States